CLINICAL TRIAL: NCT01401023
Title: Pharmacokinetics and Safety of Tigecycline in the Treatment of Clostridium Difficile Associated Diarrhea (CDAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary E. Stein, Pharm.D. (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Gary E. Stein, Pharm.D., Professor of Medicine and Pharmacology, Michigan State University
Organization: Michigan State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS1481739
Record Dates: First submitted 2011-06-16; First posted 2011-07-25 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Diarrhea; Clostridium Difficile
MeSH Terms: conditions — Diarrhea | interventions — Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clostridium difficile Patient (Experimental): Open non-comparative trial
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Tigecycline — : Standard treatment doses of oral antibiotics (vancomycin or metronidazole) for CDAD along with IV tigecycline (100 milligram loading dose followed by 50 milligrams every 12 hours) will be given to patients during their hospitalization (usually 7-14 days). Patients well enough to go home will receive only oral therapy.
  Other Names: Tygacil

SUMMARY:
This is a prospective, non-comparative, interventional, observational pilot study of the safety and pharmacokinetics of intravenous (IV) tigecycline in conjunction with standard oral therapy in patients with known mild to severe confirmed Clostridium difficile associated diarrhea (CDAD).

DETAILED DESCRIPTION:
The intervention is adding Tigecycline (standard doses) to standard oral therapy for CDAD. Patients will then be observed for clinical outcomes and relapse of CDAD.

ELIGIBILITY:
Inclusion Criteria:

* non pregnant adults (≥18 years old) with a diagnosis of mild to severe CDAD (initial or recurrent) by positive C. difficile toxin assay along with clinical symptoms (watery stools, fever, abdominal pain). Patients will receive a minimum of 3 days of tigecycline.

Exclusion Criteria:

* pregnant patients
* allergy to tetracycline (or tigecycline) antibiotics or patients with life-threatening illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Stein, PharmD, Principal Investigator — Michigan State University
Locations (2):
- United States (2):
  - Michigan State University, East Lansing, Michigan
  - Sparrow Hosptial, Lansing, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were inpatients (Sparrow Hospital) with Clostridium difficile who were treated with tigecycline. Referral base was infectious disease consultations. The first patient was enrolled 11-23-2011 and the last 9-13-2012.
Groups:
- Clostridium Difficile Patient: Open non-comparative trial
  Tygacil : : Standard treatment doses of oral antibiotics (vancomycin or metronidazole) for CDAD along with IV tigecycline (100 mg LD followed by 50 mg Q12h) will be given to patients during their hospitalization (usually 7-14 days). Patients well enough to go home will receive only oral therapy.
Period: Overall Study
Arm/Group | Clostridium Difficile Patient
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CDAD Patient: Open non-comparative trial
  Tygacil : : Standard treatment doses of oral antibiotics (vancomycin or metronidazole) for CDAD along with IV tigecycline (100 mg LD followed by 50 mg Q12h) will be given to patients during their hospitalization (usually 7-14 days). Patients well enough to go home will receive only oral therapy.
Arm/Group | CDAD Patient
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Tigecycline Along With Standard Treatments for Clostridium Difficile
Description: Serum levels of tigecycline
Time Frame: day 3 of treatment
Measure: Mean (Standard Deviation); unit: milligrams/liter
Arm/Group | Clostridium Difficile Patient
Number analyzed (Participants) | 10
milligrams/liter | 0.18 (0.14)

2. Primary Outcome: Mean (SD) Minimun Inhibitory Concentration of Tigecycline of Clostridium Difficile Isolates
Time Frame: day 1 stool sample
Measure: Mean (Standard Deviation); unit: milligram/liter
Arm/Group | Clostridium Difficile Patient
Number analyzed (Participants) | 10
milligram/liter | 0.15 (0.06)

3. Primary Outcome: Mean (SD) Serum Tigecycline Concentration Level
Description: Blood samples were obtained from each patient at the end of a dosing interval (trough concentration) on day 3 of tigecycline therapy. Serum concentrations were determined with the use of a validated high-performance liquid chromatography assay.
Time Frame: day 3 of tigecycline therapy
Measure: Mean (Standard Deviation); unit: milligram/liter
Arm/Group | Clostridium Difficile Patient
Number analyzed (Participants) | 10
milligram/liter | 0.18 (0.14)

4. Primary Outcome: Mean (SD) Stool Tigecycline Concentration Level
Description: Fecal samples were obtained from each patient at the end of a dosing interval (trough concentration) on day 3 of tigecycline therapy. Fecal concentrations were determined with the use of a validated high-performance liquid chromatography assay
Time Frame: day 3 of tigecycline therapy
Measure: Mean (Standard Deviation); unit: micrograms/gram
Arm/Group | Clostridium Difficile Patient
Number analyzed (Participants) | 10
micrograms/gram | 17.8 (23.8)

5. Primary Outcome: Pharmacokinetics of Tigecycline Along With Standard Treatments for Clostridium Difficile
Description: Stool levels of tigecycline
Time Frame: day 3 of treatment
Measure: Mean (Standard Deviation); unit: micrograms/gram
Groups:
- Clostridium Difficile Patient: Open non comparative trial
Arm/Group | Clostridium Difficile Patient
Number analyzed (Participants) | 10
micrograms/gram | 17.8 (23.8)

ADVERSE EVENTS:
Arm/Group | CDAD Patient
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDAD Patient (N=10)
Recurrence of Clostridium difficile infection (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDAD Patient (N=10)
Nausea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No